CLINICAL TRIAL: NCT04024566
Title: Aortic Stenosis Screening Using the Avicena Vivio System
Brief Title: Rapid Non-invasive Detection of Aortic Stenosis
Status: Withdrawn | Type: Observational
Why Stopped: Company changed strategic direction in Oct 2019 (staff changes; no one at company who participated in this study
Sponsor: Avicena LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AS20192
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-07

CONDITIONS: Heart Valve Diseases; Aortic Valve Disease; Heart Murmurs
Keywords: echocardiography
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Disease; Heart Murmurs

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vivio System — Optical/sensor tonometer applied to the neck over the carotid pulse (bilateral)

SUMMARY:
Avicena is developing new non-invasive methods (hardware and software) for diagnosis of a variety of heart conditions. This study is designed to compare data obtained using Avicena's device, the Vivio, to data obtained from transthoracic echocardiography (TTE) for the diagnosis of moderate-to-severe aortic stenosis. Aortic stenosis (AS) is a disease of the valve (aortic valve) that separates the left ventricle of the heart from the aorta. When AS is severe, the heart cannot pump adequate amounts of blood into the arterial tree. AS is often silent until the disease is severe. This study compares a rapid test using Vivio to a longer and more expensive test that is the current gold standard for diagnosis of AS, TTE.

DETAILED DESCRIPTION:
The study proposed here is a research study to develop the Vivio system for diagnosis of severe AS. The data gathered in this study will be used to optimize the Avicena software algorithm used to make the diagnosis of AS.

The Vivio device is an optical-type tonometer that operates based on capturing the vibrations of the skin due to the arterial pulse pressure wave as it propagates through the underlying carotid vessel. When applied to the neck over the subject's carotid pulse, an arterial waveform (pressure tracing) and heart sounds are sensed, and sent to an iPad using Bluetooth, then sent to Avicena for analysis.

After informed consent subjects will undergo a brief cardiac-focused history and examination. All subjects will have bilateral exams with the Vivio (~5 minutes each) conducted by a study doctor or nurse, and a standard clinical resting TTE conducted by a certified technician. The entire study visit should take 1.5 hours, and there is no follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects >60 years of age
2. Ability to understand and sign informed consent
3. Willingness to undergo study protocol (in Pasadena CA)

Exclusion Criteria:

1. Inability to provide informed consent
2. History of carotid sinus hypersensitivity (fainting in response to minimal touching or positioning of the neck)
3. History of significant or symptomatic carotid artery disease, or carotid artery stenting or surgery
4. History of aortic valve surgery or transcatheter aortic valve replacement
5. Absent carotid pulse on initial examination (inability to palpate the carotid pulse)
6. Open skin lesions at the site of Vivio application/examination
7. Presence of a carotid bruit on examination

Ages: 60 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe, symptomatic AS incidence increases with age, so that most patients do not experience symptoms until after age 60. For this reason, to enrich for the population of patients with potential AS, subjects over age 65 will be studied.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Optimized algorithm for diagnosis of AS | 2 years
  Data collected in this study will be analyzed by multiple mathematical approaches to develop an optimized algorithm for detection of severe AS

SECONDARY OUTCOMES:
Positive predictive value (PPV) of Vivio in the diagnosis of severe AS | 2 years
  PPV for detecting AS by Vivio compared to PPV for 2D TTE

CONTACTS AND LOCATIONS:
Overall Officials: Sean Brady, JD, Study Director — Chief Executive Officer
Locations (1):
- Avicena, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed AK, Garberich R, Gossl M, Tindell L, Williams K, Dennis S, Bae R, Soraja P. A novel method of non-invasive screening for patients with aortic stenosis. JACC March 12, 2019, 73 (9 Supplement 1) 1995; DOI:10.1016/S0735-1097(19)32601-4